CLINICAL TRIAL: NCT02949648
Title: A Pilot Study on Electronic Cigarette Use and Their Impact on Smoking and Quitting in Youth
Brief Title: Electronic Cigarette Use and Quitting in Youth
Status: Completed | Type: Observational
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Wang Man-Ping, Assisstant Professor, The University of Hong Kong
Other Study IDs: EC use and quitting in youth
Record Dates: First submitted 2016-05-19; First posted 2016-10-31 (Estimated); Last update posted 2016-10-31 (Estimated); Status verified 2016-10

CONDITIONS: Smoking
Keywords: Electronic cigarette
MeSH Terms: conditions — Smoking; Vaping

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Electronic cigarette ever user: Youth Quitline callers who reported ever use of e-cigarette at baseline.
  Interventions: Device: Electronic cigarette
- Electronic cigarette never user: Youth Quitline callers who reported never use of e-cigarette at baseline.

INTERVENTIONS:
Device: Electronic cigarette — Electronic cigarettes are devices that do not burn or use tobacco leaves but instead vaporize a solution the user then inhales. The device contains an electronic vaporization system, rechargeable batteries, electronic controls and cartridges of the liquid is vaporized.
  Other Names: Electronic nicotine delivery system
  Groups: Electronic cigarette ever user

SUMMARY:
A mixed method (longitudinal, trajectory and qualitative studies) to provide comprehensive evidence on the impact of e-cigarette use on smoking and quitting among smoking youth in Hong Kong.

DETAILED DESCRIPTION:
Subjects are from a cohort of Youth Quitline callers and smoking youth (N=200) in Hong Kong. The longitudinal study will investigate the effects of baseline e-cigarette use on quitting (including relapse), nicotine addiction and intention to smoke at 12-month telephone follow-up. A qualitative study will be conducted on 10 ex- and 10 current smokers to supplement and facilitate interpretation of the quantitative findings.

ELIGIBILITY:
Inclusion Criteria:

1. Ethnic Chinese
2. Cantonese speakers
3. Smoke at least 1 cigarette in the past 30 days

Exclusion Criteria:

1. Psychologically or physically unable to communicate
2. Undergoing other smoking cessation programme

Max Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Youth in Hong Kong
Sampling Method: Non-Probability Sample
Enrollment: 189 (Actual)
Dates: Start 2015-09; Primary Completion 2016-06 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
7-day point prevalence abstinence assessed in the telephone follow-up survey | 12 months after baseline survey
  Self-reported 7-day point prevalence abstinence (PPA) is a validated, commonly used measure of smoking cessation. Subjects who reports no smoking in the preceding 7 days at the time of 12-month survey in the follow-up are regarded as quitters.
  This measure has serval advantages compared to continuous abstinence. First, it can include smokers who take delayed action and quit. It also allows relapses to occur in the follow up period, without classifying smokers as permanent failure. Third, it does not rely on recall of past events happened long ago.

SECONDARY OUTCOMES:
Quit attempts assessed in the telephone follow-up survey | 12 months after baseline survey
  Smokers report how many times they try to abstain from cigarette for more than 24 hours in the whole follow-up period
Intention to quit assessed in the telephone follow-up survey | 12 months after baseline survey
  Smokers report whether they intend to quit smoking at the time of 12-month survey in the follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Man Ping Wang, PhD, Principal Investigator — mpwang@hku.hk
Locations (1):
- Youth Quitline, School of Nursing, The University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No